CLINICAL TRIAL: NCT01870544
Title: Does Weight Loss Surgery and Probiotic Supplementation Lead to a "Lean" Gut Microbiota?
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tufts Obesity Study
Record Dates: First submitted 2013-05-13; First posted 2013-06-06 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
Keywords: gastric bypass; microbiota; probiotic
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LGG Administration (Experimental): Lactobacillus Rhamnosus GG (LGG) will be taken orally for 44 days. The daily dose is 2*10^10 organisms. The LGG is contained in capsules (1*10^10 organisms per capsule), and two capsules will be taken per day.
  Interventions: Dietary Supplement: Lactobacillus Rhamnosus GG
- Placebo (Placebo Comparator): Placebo to be taken orally for 44 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus Rhamnosus GG — LGG will be administered orally for 44 days
  Arms: LGG Administration
Dietary Supplement: Placebo — placebo will be administered daily for 44 days
  Arms: Placebo

SUMMARY:
The purpose of the weight-loss study is to characterize the effect of LGG supplementation on the relative abundance of phyla in the gut microbiota of patients undergoing gastric bypass and sleeve gastrectomy surgery, and to elucidate a relationship between the gut microbiota pattern and the degree of weight-loss post-surgery.

The investigators hypothesize that LGG administration will result in a "leaner" pattern of gut microbiota that will lead to higher weight loss at 3 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Able to give informed consent and report on side effects
3. Tolerating an oral/enteral diet
4. Stable comorbid conditions
5. Outpatient

Exclusion Criteria:

1. Inpatients
2. Pregnancy (urine test done on all patients routinely pre-op)/ unwilling to comply with contraceptive requirement after gastric bypass surgery
3. Known use of LGG or another probiotic (not including yogurt) within the previous 30 days
4. Presence of an active bowel leak, acute abdomen, active intestinal disease, or significant bowel dysfunction
5. Presence of an absolute neutrophil count less than 500 per cubic mm (must have had a Complete Blood Count within the last 6 months) or anticipation post chemotherapy that the absolute neutrophil count will fall below 500 per cubic mm.
6. History of adverse reaction to product containing lactobacillus
7. Active colitis (*see definition below)
8. Known or suspected allergies to probiotics, lactobacillus, milk protein, or microcrystalline cellulose
9. Structural heart disease, history of endocarditis or valve replacement, implanted cardiac device, congestive heart failure
10. Positive baseline stool culture for LGG
11. Recent or planned chemotherapy or radiation therapy
12. Solid organ transplant within the prior year
13. Stem cell transplant within the prior year
14. On active immunosuppressive medication [anti-rejection, injectable immunosuppressive drugs for autoimmune disease, or corticosteroids (greater than ½ mg per kg body weight of prednisone or its equivalent) not including inhaled or topical steroids]
15. Allergy or intolerance to or contraindication to two or more of the rescue antibiotic regimens (ampicillin, clindamycin, moxifloxacin)
16. Participating in another clinical trial
17. Uncontrolled psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 4 months

SECONDARY OUTCOMES:
Percentage of Bacteria Phyla | 4 months
  We will specifically look at the percentages of different bacterial phyla in the stool and intestine

CONTACTS AND LOCATIONS:
Overall Officials: Shira Doron, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center Weight and Wellness Center, Boston, Massachusetts, United States